CLINICAL TRIAL: NCT03201302
Title: The KOMOtini BONE Study: Evaluation of Sports-Related Osteogenic Potential in School-Aged Children
Brief Title: The KOMOtini BONE Study: Evaluation of the Osteogenic Potential of Sports
Acronym: KOMO-BONE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ioannis G. Fatouros (Other)
Collaborators: Democritus University of Thrace (Other)
Responsible Party: Sponsor-Investigator, Ioannis G. Fatouros, Associate Professor, University of Thessaly
Organization: University of Thessaly (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DUTH-UTH
Record Dates: First submitted 2017-01-02; First posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Bone Mineral Content; Bone Density; Bone Turnover Markers; Athletic Performance
Keywords: bone; childhood; pre-adolescence; bone turnover markers; sclerostin; sports; physical activity; nutrition
MeSH Terms: conditions — Sclerosteosis; Motor Activity | interventions — Stair Climbing; Swimming

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (16):
- School physical education class (Experimental): Children who participated only in their school physical activity classes only for the entire school year.
  Interventions: Other: School physical education class
- Taekwondo (Experimental): Children who participated in organized Taekwondo training for the entire school year.
  Interventions: Other: Taekwondo
- Martial arts (Experimental): Children who participated in organized Martial arts training for the entire school year.
  Interventions: Other: Martial arts
- Climbing (Experimental): Children who participated in organized climbing training for the entire school year.
  Interventions: Other: Climbing
- Volleyball (Experimental): Children who participated in organized volleyball training for the entire school year.
  Interventions: Other: Volleyball
- Artistic gymnastics (Experimental): Children who participated in organized artistic gymnastics training for the entire school year.
  Interventions: Other: Artistic gymnastics
- Swimming (Experimental): Children who participated in organized swimming training for the entire school year.
  Interventions: Other: Swimming
- Dance (Experimental): Children who participated in organized dance training for the entire school year.
  Interventions: Other: Dance
- Basketball (Experimental): Children who participated in organized basketball training for the entire school year.
  Interventions: Other: Basketball
- Wrestling (Experimental): Children who participated in organized wrestling training for the entire school year.
  Interventions: Other: Wrestling
- Football (soccer) (Experimental): Children who participated in organized football (soccer) training for the entire school year.
  Interventions: Other: Football (soccer)
- Rhythmic gymnastics (Experimental): Children who participated in organized rhythmic gymnastics training for the entire school year.
  Interventions: Other: Rhythmic gymnastics
- Track and field (Experimental): Children who participated in organized track and field training for the entire school year.
  Interventions: Other: Track and field
- Tennis (Experimental): Children who participated in organized tennis training for the entire school year.
  Interventions: Other: Tennis
- Combination of activities 1 (Experimental): Children who participated in two different weight-bearing activities for the entire school year.
  Interventions: Other: Combination of activities 1
- Combination of activities 2 (Experimental): Children who participated in one weight-bearing and in one non weight-bearing activity for the entire school year.
  Interventions: Other: Combination of activities 2

INTERVENTIONS:
Other: School physical education class — Children participated only in school physical education classes only.
  Arms: School physical education class
Other: Taekwondo — Children participated only in taekwondo training only.
  Arms: Taekwondo
Other: Martial arts — Children participated only in martial arts training only.
  Arms: Martial arts
Other: Climbing — Children participated only in climbing training only.
  Arms: Climbing
Other: Volleyball — Children participated only in volleyball training only.
  Arms: Volleyball
Other: Artistic gymnastics — Children participated only in artistic gymnastics training only.
  Arms: Artistic gymnastics
Other: Swimming — Children participated only in swimming training only.
  Arms: Swimming
Other: Dance — Children participated only in dance training only.
  Arms: Dance
Other: Basketball — Children participated only in basketball training only.
  Arms: Basketball
Other: Wrestling — Children participated only in wrestling training only.
  Arms: Wrestling
Other: Football (soccer) — Children participated only in football (soccer) training only.
  Arms: Football (soccer)
Other: Rhythmic gymnastics — Children participated only in rhythmic gymnastics training only.
  Arms: Rhythmic gymnastics
Other: Track and field — Children participated only in track and field training only.
  Arms: Track and field
Other: Tennis — Children participated only in tennis training only.
  Arms: Tennis
Other: Combination of activities 1 — Children participated in two weight-bearing activities.
  Arms: Combination of activities 1
Other: Combination of activities 2 — Children participated in one weight-bearing activity and in one non weight-bearing activity.
  Arms: Combination of activities 2

SUMMARY:
Bone mass develops throughout childhood and adolescence until a peak bone mass is achieved during early adulthood. Fracture risk later in life can be predicted at a large extent by peak bone mass. Occurence of sarcopenia and osteoporosis (i.e. loss of mone mass) during late adulthood has been strongly associated with the degree of bone mineralization during early life. Nearly 50% of total bone mineral content (BMC) reached during adulthood is obtained during pre-adolescence rendering this period critical for skeletal health and is considered as an optimal period for bone/skeletal growth since during this time bones are more adaptable to osteogenic stimuli such as exercise-induced mechanical loading. Organized sport activities and/or nutrition appear to affect profoundly bone mineral density (BMD), BMC, bone geometry, and overall skeletal health during preadolescence offering an effective type of prevention of osteoporosis, a condition very difficult to treat later in life. Evidence suggest that some modes of exercise activities may be more effective (osteogenic) for bone development due to the magnitude and type of mechanical strain placed on long bones causing them to be more dense. Weight-bearing activities (e.g. running, jumping etc.) are believed to be more osteogenic than non-weight bearing activities. However, more research is required in order to determine: i) whether weight-bearing activities are more osteogenic than non weight -bearing activities during childhood and ii) the osteogenic potential of a large number of sport activities used by school-children as compared to a control treatment of no participation in organized sport activities. The present trial attempted to compare a large number of different sport activities in respect to their osteogenic potential based on training variables that are thought to affect osteogenesis while at the same time allows direct comparison of exercise modes that are entirely different. Therefore, the goal of this investigation was to determine the osteogenic potential of a large number of exercise training activities in boys and girls of 8-12 years of age during an entire primary school season.

DETAILED DESCRIPTION:
Healthy, previously untrained, pre-pubertal boys and girls (N=335) were assigned to 16 different groups: 1) physical education, i.e. children participated only school in physical education classes (control group), 2) football (soccer) training, 3) basketball training, 4) volleyball training, 5) wrestling training, 6) martial arts training, 7) tennis training, 8) track and field training, 9) taekwondo training, 10) rhythmic gymnastics training, 11) artistic gymnastics training, 12) dance training, 13) swimming training, 14) climbing training, 15) two weight-bearing training modes, and 16) one weight-bearing and one non-weight bearing activity. Exercise training was performed three times per week for nine months and each training session had a 60-minute duration (except for the physical education classes at school in the control group). Anthropometric measurements (body height, body mass, and length and circumferences of various body segments), blood sampling, measurements of body composition (using dual X-ray energy absorptiometry or DEXA and skinfold calibers), bone measurements (bone density and bone mineral content at lumbar spine, both hips, both wrists and whole body using DEXA), and performance (cardiorespiratory fitness, muscle strength, muscle power, flexibility and motor ability) were performed at baseline and after the completion of a 9-month training intervention. Nutritional intake and habitual physical activity were measured at baseline, mid-training and post-training (using diet recalls and accelerometry, respectively). Intensity and volume of training was measured once every three months using heart rate monitoring, accelerometry, Global Positioning System (GPS) devices and jump measurement. Furthermore, two other studies were also performed as a part of this project: a) assessment of physical activity during physical education classes for primary school (using accelerometry, GPS instrumentation and jump measurement) and b) a smaller number of participants in the football, track and field, swimming and tennis training groups provided blood samples before and after a training session at baseline.

ELIGIBILITY:
Inclusion criteria

* were 8-12 years and pre-pubertal
* were healthy and had no prior bone fractures or related surgical operation
* had not been involved in organized sport activities previously
* their body fat was <30%, e) had no history of growth irregularities
* were not receiving agents or drugs that affect bone tissue (e.g. Gonadotropin-Releasing Hormone (GnRH) agonists, antiresorptive, bisphosphonates, etc.)

Exclusion Criteria:

* had prior bone fractures or related surgical operation
* had been involved in organized sport activities previously
* their body fat was >30%
* had history of growth irregularities
* were receiving agents or drugs that affect bone tissue (e.g. GnRH agonists, antiresorptive, bisphosphonates, etc.)
* missed more than 10% of training sessions

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 335 (Actual)
Dates: Start 2013-04; Primary Completion 2014-06 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Changes in bone mineral content | At baseline and 9 months.
  Using a whole body, hip (left and right), lumbar spine, and wrist (left and right) scans performed by a dual-energy x-ray absorptiometry scanner.
Changes in bone density | At baseline and 9 months.
  Using a whole body, hip (left and right), lumbar spine, and wrist (left and right) scans performed by a dual-energy x-ray absorptiometry scanner.
Changes in area of different regions and sub-regions | At baseline and 9 months.
  Using a whole body, hip (left and right), lumbar spine, and wrist (left and right) scans performed by a dual-energy x-ray absorptiometry scanner.
Changes in bone resorption | At baseline and 9 months.
  By measuring blood levels of sclerostin, calcium, phosphorus, magnesium, creatinine, alkaline phosphatase (ALP), vitamin D (if budget allows), serum procollagen type 1 aminoterminal propeptide (P1NP, if budget allows) and isomer of the Carboxy-terminal telopeptide of type 1 collagen (CTX-1, if budget allows).
Changes in cardiorespiratory performance | At baseline and 9 months.
  Using a shuttle run test
Changes in muscle power performance of the lower limbs | At baseline and 9 months.
  Using long jump test, standing long jump test, countermovement jump test and the Abalakov jump.
Changes in flexibility performance | At baseline and 9 months.
  Using the sit and reach test
Changes in muscle strength | At baseline and immediately after the completion of training.
  Using handgrip dynamometry (left and right arm)
Changes in motor performance | At baseline and 9 months.
  Using a standard motor ability test battery
Changes in stature (cm) | At baseline and 9 months.
Changes in seated height (cm) | At baseline and 9 months.
Changes in body mass (kg) | At baseline and 9 months.
Changes in body mass index (BMI) | At baseline and 9 months.
  Calculated as body mass (kg) divided by the height (m) squared.
Changes in arm span | At baseline and 9 months.
Changes in tibia length | At baseline and 9 months.
Changes in biacromial length | At baseline and 9 months.
Changes in chest width | At baseline and 9 months.
Changes in waist circumference | At baseline and 9 months.
Changes in hip circumference | At baseline and 9 months.
Changes in forearm length | At baseline and 9 months.
Changes in hand length | At baseline and 9 months.
Changes in body fat mass | At baseline and 9 months.
  Body composition was measured using a dual-energy x-ray absorptiometry scanner (DEXA). DEXA instrumentation allowed the measurement of regional (legs, arms, trunk) weight, body fat (%), and fat mass (kg).
Changes in lean body mass | At baseline and 9 months.
  Body composition was measured using a dual-energy x-ray absorptiometry scanner (DEXA). DEXA instrumentation allowed the measurement of regional (legs, arms) weight, lean mass (kg).

SECONDARY OUTCOMES:
Changes in sexual maturation | At baseline and 9 months.
  Sexual maturation was assessed using the Tanner scale with stages of sexual maturation, orchidometer for boys. Potentially sexual maturation will be assessed also using measurement of hormonal concentration in the blood (if budget allows).
Changes in diet intake | At baseline, after 4,5 months of training and after 9 months of training.
  Food intake was measured using diet recalls. Participants and their parents were instructed how to record the type and the quantity of solid and liquid foods consumed daily. Daily caloric intake as well daily intake of all nutrients was estimated using a nutritional software.
Changes in habitual physical activity | At baseline, after 4,5 months of training and after 9 months of training.
  Daily habitual physical activity was measured using an accelerometer.
Changes in training intensity | At baseline, after 4,5 months of training and after 9 months of training.
  Training intensity was measured in two consecutive training sessions for each sport activity at three time points during the intervention. Training intensity was assessed using the following: a) heart rate responses using heart rate monitors, b) accelerometry (except for swimming), c) GPS instrumentation (global positioning system) for outdoor activities only.
Changes in training volume | At baseline, after 4,5 months of training and after 9 months of training.
  Training volume was measured in two consecutive training sessions for each sport activity at three time points during the intervention. Training volume was measured using the following: a) total distance covered using GPS instrumentation and accelerometry for outdoor activities, b) accelerometry for indoor activities, c) recording of total meters covered during a session for swimming and d) total vertical jump number.

CONTACTS AND LOCATIONS:
Overall Officials: Antonis Kambas, Study Director — Democritus University of Thrace; Diamanda Leontsini, Principal Investigator — Democritus University of Thrace
Locations (1):
- Laboratory of Physical Education and Sports, Democritus University of Thrace, School of Physical Education & Sports Sciences, Komotini, Greece

IPD SHARING:
Plan to Share IPD: No